CLINICAL TRIAL: NCT06372535
Title: Dose-Response Effects of Tai Chi Chuan Interventions on Cognitive Function in Mild Cognitive Impairment
Brief Title: Effects of Tai Chi Chuan With Different Doses on Cognitive Function in Elderly Patients With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lidian Chen (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor-Investigator, Lidian Chen, PhD, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FujianUTCM-1
Record Dates: First submitted 2024-03-18; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Tai Chi Chuan; Cognitive Function; Dose-response
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Tai Chi Chuan Group1 (Experimental): Tai Chi Chuan 0.5 hour/session, 5 sessions/week for 8 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 1）
- Tai Chi Chuan Group2 (Experimental): Tai Chi Chuan 0.5 hour/session, 5 sessions/week for 16 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 2）
- Tai Chi Chuan Group3 (Experimental): Tai Chi Chuan 0.5 hour/session, 5 sessions/week for 24 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 3）
- Tai Chi Chuan Group4 (Experimental): Tai Chi Chuan 1 hour/session, 5 sessions/week for 8 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 4）
- Tai Chi Chuan Group5 (Experimental): Tai Chi Chuan 1 hour/session, 5 sessions/week for 16 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 5）
- Tai Chi Chuan Group6 (Experimental): Tai Chi Chuan 1 hour/session, 5 sessions/week for 24 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 6）
- Tai Chi Chuan Group7 (Experimental): Tai Chi Chuan 1.5 hour/session, 5 sessions/week for 8 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 7）
- Tai Chi Chuan Group8 (Experimental): Tai Chi Chuan 1.5 hour/session, 5 sessions/week for 16 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 8）
- Tai Chi Chuan Group9 (Experimental): Tai Chi Chuan 1.5 hour/session, 5 sessions/week for 24 weeks.
  Interventions: Behavioral: Tai Chi Chuan （dose 9）

INTERVENTIONS:
Behavioral: Tai Chi Chuan （dose 1） — Participants would take 24-form simplified Tai Chi Chuan 0.5 hour/session, 5 sessions/week for 8 weeks.
  There were 10 minutes warm-up, 30 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group1
Behavioral: Tai Chi Chuan （dose 2） — Participants would take 24-form simplified Tai Chi Chuan 0.5 hour/session, 5 sessions/week for 16 weeks.
  There were 10 minutes warm-up, 30 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group2
Behavioral: Tai Chi Chuan （dose 3） — Participants would take 24-form simplified Tai Chi Chuan 0.5 hour/session, 5 sessions/week for 24 weeks.
  There were 10 minutes warm-up, 30 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group3
Behavioral: Tai Chi Chuan （dose 4） — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 5 sessions/week for 8 weeks.
  There were 10 minutes warm-up, 60 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group4
Behavioral: Tai Chi Chuan （dose 5） — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 5 sessions/week for 16 weeks.
  There were 10 minutes warm-up, 60 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group5
Behavioral: Tai Chi Chuan （dose 6） — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 5 sessions/week for 24 weeks.
  There were 10 minutes warm-up, 60 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group6
Behavioral: Tai Chi Chuan （dose 7） — Participants would take 24-form simplified Tai Chi Chuan 1.5 hour/session, 5 sessions/week for 8 weeks.
  There were 10 minutes warm-up, 90 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group7
Behavioral: Tai Chi Chuan （dose 8） — Participants would take 24-form simplified Tai Chi Chuan 1.5 hour/session, 5 sessions/week for 16 weeks.
  There were 10 minutes warm-up, 90 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group8
Behavioral: Tai Chi Chuan （dose 9） — Participants would take 24-form simplified Tai Chi Chuan 1.5 hour/session, 5 sessions/week for 24 weeks.
  There were 10 minutes warm-up, 90 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training.
  Arms: Tai Chi Chuan Group9

SUMMARY:
To determine the impact of Tai Chi Chuan with different exercise volume on cognitive function in elderly patients with mild cognitive impairment.

DETAILED DESCRIPTION:
Taking MCI as a potential gateway, early intervention to delay the occurrence of dementia has become an important consensus in this field. Exercise is an important means to improve cognitive function in MCI, but the effect of exercise is influenced by the dosage. Tai Chi Chuan, is a moderate intensity aerobic exercise. Previous studies by our team and others had confirmed its effect on cognitive function in MCI. However, the dose parameters of Tai Chi Chuan exercise varied in these studies, and the dose-response relationship is still unclear. The purpose of this study is to explore the dose-response relationship between different volume of Tai Chi Chuan exercise and cognitive function（global cognition and cognition of subdomains）in elderly MCI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of mild cognitive impairment, not demented;
2. Age ≥ 60 years old;
3. Informed consent and voluntary participation.

Exclusion Criteria:

1. Geriatric Depression Scale score ≥ 9 points
2. Cognitive impairment caused by other reasons, taking drugs, poisoning, etc;
3. Suffer from severe musculoskeletal system diseases and other contraindications to exercise and are not suitable for Tai Chi training, such as those who suffer from stroke, Parkinson's disease, and have a history of lower limb arthritis, hip and knee joint replacement, etc;
4. Patients with severe heart, liver, kidney failure, malignant tumors, and other major diseases;
5. Individuals with visual/auditory impairments, writing/reading impairments, illiteracy, etc. that affect training and evaluation;
6. Individuals with uncontrolled hypertension (systolic blood pressure greater than 160mmHg or diastolic blood pressure greater than 100mmHg after medication);
7. Participating in other experiments that influence this study;
8. Engaged in regular exercise in the last three months (at least 3 times a week, at least 20 minutes of regular exercise each time.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 8 weeks, 16 weeks, 24 weeks
  Global cognition

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | 52 weeks
  Global cognition
Wechsler Memory Scale | 8 weeks[the duration of intervention arm greater than or equal 8 weeks], 16 weeks [the duration of intervention arm greater than or equal 16 weeks], 24 weeks [the duration of intervention arm is 24 weeks] and 52 weeks
  Memory function
Digital Symbol test | 8 weeks[the duration of intervention arm greater than or equal 8 weeks], 16 weeks [the duration of intervention arm greater than or equal 16 weeks], 24 weeks [the duration of intervention arm is 24 weeks] and 52 weeks
  Attention
Trial Making Test part B | 8 weeks[the duration of intervention arm greater than or equal 8 weeks], 16 weeks [the duration of intervention arm greater than or equal 16 weeks], 24 weeks [the duration of intervention arm is 24 weeks] and 52 weeks
  Executive function
Stroop color word test | 8 weeks[the duration of intervention arm greater than or equal 8 weeks], 16 weeks [the duration of intervention arm greater than or equal 16 weeks], 24 weeks [the duration of intervention arm is 24 weeks] and 52 weeks
  Processing speed
Boston naming test | 8 weeks[the duration of intervention arm greater than or equal 8 weeks], 16 weeks [the duration of intervention arm greater than or equal 16 weeks], 24 weeks [the duration of intervention arm is 24 weeks] and 52 weeks
  Verbal fluency
Rey-Osterrieth complex graphics test | 8 weeks[the duration of intervention arm greater than or equal 8 weeks], 16 weeks [the duration of intervention arm greater than or equal 16 weeks], 24 weeks [the duration of intervention arm is 24 weeks] and 52 weeks
  Rey-Osterrieth complex graphics test
Rey Auditory Verbal Learning Test | 8 weeks[the duration of intervention arm greater than or equal 8 weeks], 16 weeks [the duration of intervention arm greater than or equal 16 weeks], 24 weeks [the duration of intervention arm is 24 weeks] and 52 weeks
  Episodic memory

OTHER OUTCOMES:
Blood glucose metabolism index | 8 weeks or 16 weeks or 24 weeks [post-intervention] and 52weeks
  fasting blood glucose
Blood lipid metabolism index | 8 weeks or 16 weeks or 24 weeks [post-intervention] and 52weeks
  total cholesterol (TC), total triglyceride (TG), low density lipoprotein (LDL), high density lipoprotein (HDL)
Functional Magnetic Resonance Imaging | 8 weeks or 16 weeks or 24 weeks [post-intervention]
  Functional Magnetic Resonance Imaging
Electroencephalogram | 8 weeks or 16 weeks or 24 weeks [post-intervention]
  1. Resting-State Electroencephalogram (EEG) Power Spectrum Changes. The power spectrum density of the brain in a relaxed state is measured using a resting-state electroencephalogram (EEG) for the delta (1-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and gamma (30-100 Hz) bands. Changes in the power of these frequency bands before and after the intervention are assessed to reflect changes in the level of brain activity.
  2. Task-Related Brain Electrophysiological Activity While performing specific cognitive tasks, brain activity is recorded using an Electroencephalogram (EEG), and task-related EEG event-related potentials are analyzed.
Heart rate variability | 8 weeks or 16 weeks or 24 weeks [post-intervention]
  cardiac autonomic modulations
Gut microflora | 8 weeks or 16 weeks or 24 weeks [post-intervention] and 52weeks
  16S rRNA amplification sequencing will be used to detect intestinal microbiota. Stool sample from each sub center will be stored within 1 h of collection at - 80 °C freezer. Subsequently, the fecal samples will be stored in dry ice and transported in batches to the laboratory within 8 hours, followed by storage in - 80 °C freezer.
Sleep Quality | 8 weeks or 16 weeks or 24 weeks [post-intervention] and 52weeks
  The Pittsburgh Sleep Quality Index will be used to evaluate sleep quality, with a total score of 0-21. The higher the score, the poorer the sleep quality.
General health | 8 weeks or 16 weeks or 24 weeks [post-intervention] and 52weeks
  12-Item Short Form Health Survey will be used to evaluate general health. the higher the total score, the better the individual's health status.